CLINICAL TRIAL: NCT04011696
Title: Monofocal Extended Range of Vision (MERoV) Study
Acronym: MERoV
Status: Completed | Type: Observational
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Collaborators: King's College London (Other); European Society of Cataract and Refractive Surgeons (Other)
Responsible Party: Sponsor
Other Study IDs: 264296
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Pseudophakia; Accomodation; Aberration, Corneal Wavefront
Keywords: pseudoaccommodation; monofocal IOL; cataract surgery
MeSH Terms: conditions — Pseudophakia; Corneal Wavefront Aberration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators are proposing this research project to:

1. Screen a set of patients after normal cataract surgery with a single focus lens aimed at good distance vision at 3 months after surgery to identify patients who are able to see and read well without glasses.
2. Identify the combination of factors responsible for this phenomenon in the patients who are achieving this.

Potentially eligible patients will be given an invitation letter and patient information sheet on the day they arrive for surgery. They will then be asked if they are happy to be contacted by phone 2-4 weeks post-surgery with a view to booking them into an additional research visit at 3 months after their surgery. At 3 months after surgery they will have their un-corrected vision checked. They will also have their reading speed assessed without any glasses. They will undergo a through refractive check by an optometrist to assess the power of the spectacles (if needed) and following this they will have a scan of the eye (a technique known as wave front analysis which uses very sophisticated optics) to capture the optical distortions in the structures of the eye.

If this study is able identify factor/s responsible for giving good unaided reading and distance vision then this factor can be reproduced in eyes undergoing cataract surgery. This will mean that the patients can have an increased option of spectacle independence without the need for expensive multifocal IOLs and their associated side effects such as glare and halos, particularly at night.

DETAILED DESCRIPTION:
TYPE OF THE STUDY:

A prospective, non-blinded, non-randomized, single eye cohort study in patients who had uneventful cataract surgery with a monofocal IOL.

Potentially eligible patients will be given an invitation letter and patient information sheet on the day they arrive for surgery. They will then be asked if they are happy to be contacted by phone 2-4 weeks post-surgery with a view to booking them into an additional research visit at 3 months after their surgery.

Inclusion criteria

1. Uneventful cataract surgery
2. Sequential recruitment
3. Potential to see 20/40 (6/12) unaided or better postoperatively
4. No significant macular pathology
5. Willing to follow up at 3 months

Exclusion criteria

1. Patients under 20 years of age
2. Any ocular co-morbidity, which will preclude an expected postoperative 20/40 (6/12) unaided, distance vision. (e.g. amblyopia, corneal pathology, age related macular degeneration, glaucoma, diabetic retinopathy, other previous ocular surgeries)
3. Posterior capsule opacification
4. Inability to read English text or physically or mentally unable to cooperate with the postoperative assessment

At 3 months, uniocular unaided distance LogMAR acuity will be recorded. An OCT scan will be performed to establish macular integrity. Pupil size, manifest refraction, measurement of any deviations of the optical rays (called as wavefront aberrometry) will be performed using a iTrace (Tracy Technology) wavefront aberrometer. Unaided reading speed and critical print size will be measured using a Salzberg Reading Desk. Examination time per patient: 40 mins in total. Multivariate statistical analysis will be performed. Power calculation showed a need to examine 412 patients.

ELIGIBILITY:
Inclusion Criteria:

* Uneventful cataract surgery, sequential recruitment, potential to see 20/40 (6/12) unaided or better postoperatively, no significant macular pathology and willing to follow up at 3 months.

Exclusion Criteria:

* Any ocular co-morbidity, which will preclude an expected postoperative 20/40 (6/12) unaided, distance vision. (e.g. amblyopia, corneal pathology, age related macular degeneration, glaucoma, diabetic retinopathy, other previous ocular surgeries), posterior capsule opacification,inability to read English text or physically or mentally unable to and cooperate with the postoperative assessment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For the purpose of this research, the notes of all the patient undergoing routine NHS cataract surgery will be assessed by the research nurse to see if they have a potential to have 6/12 or better vision after cataract surgery. If so, they will be given an invitation letter and patient information sheet on the day they arrive for surgery. They will then be asked if they are happy to be contacted by phone 2-4 weeks post-surgery with a view to booking them into an additional research visit at 3 months after their surgery
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Uncorrected distance and near vision | 3 months postoperatively
  Uncorrected distance of 20/40 and near of J4

SECONDARY OUTCOMES:
Spherical error | 3 months postoperatively
  Spherical error on manifest refraction
astigmatic error | 3 months postoperatively
  astigmatic error on manifest refraction
Pupil size | 3 months postoperatively
  Pupil size in mesopic condition
Total spherical and vertical coma aberrations | 3 months postoperatively
  Total spherical and vertical coma aberrations on aberrometry
Reading speed and critical font size | 3 months postoperatively
  Measured on Salzburg's reading desk

CONTACTS AND LOCATIONS:
Overall Officials: Mayank A Nanavaty, FRCOphth,PhD, Study Chair — Brighton and Sussex University Hospitals NHS Trust; David J Spalton, FRCOphth, Principal Investigator — King's College London; Catey Bunce, DSc, Principal Investigator — King's College London
Locations (1):
- Mayank Nanavaty, Brighton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The data will be collected in paper files and NHS computers. No external agency will have access to the study data.

REFERENCES:
- [Background] Nanavaty MA, Vasavada AR, Patel AS, Raj SM, Desai TH. Analysis of patients with good uncorrected distance and near vision after monofocal intraocular lens implantation. J Cataract Refract Surg. 2006 Jul;32(7):1091-7. doi: 10.1016/j.jcrs.2006.03.021. PMID 16857493
- [Background] Nanavaty MA, Spalton DJ, Boyce J, Saha S, Marshall J. Wavefront aberrations, depth of focus, and contrast sensitivity with aspheric and spherical intraocular lenses: fellow-eye study. J Cataract Refract Surg. 2009 Apr;35(4):663-71. doi: 10.1016/j.jcrs.2008.12.011. PMID 19304086
- [Background] Nanavaty MA, Spalton DJ, Marshall J. Effect of intraocular lens asphericity on vertical coma aberration. J Cataract Refract Surg. 2010 Feb;36(2):215-21. doi: 10.1016/j.jcrs.2009.08.024. PMID 20152600
- [Derived] Nanavaty MA, Mukhija R, Ashena Z, Bunce C, Spalton DJ. Incidence and factors for pseudoaccommodation after monofocal lens implantation: the Monofocal Extended Range of Vision study. J Cataract Refract Surg. 2023 Dec 1;49(12):1229-1235. doi: 10.1097/j.jcrs.0000000000001302. PMID 37769187